CLINICAL TRIAL: NCT01730209
Title: Efficacy of RAD001/Everolimus in Autism and NeuroPsychological Deficits in Children With Tuberous Sclerosis Complex
Acronym: RAPIT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Utrecht University (Other)
Responsible Party: Principal Investigator, M.C.Y. de Wit, MD PhD, Pediatric Neurologist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL38619.078.11
Record Dates: First submitted 2012-10-26; First posted 2012-11-21 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Tuberous Sclerosis Complex; TSC Related Cognitive Disability; TSC Related Autism; TSC Related Learning Problems
Keywords: Tuberous Sclerosis Complex; TSC; Autism; Learning problems; Everolimus; RAD001; Treatment; Cognition; Intellectual disability
MeSH Terms: conditions — Tuberous Sclerosis; Autistic Disorder; Intellectual Disability | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (Experimental): Everolimus once daily for 1 year, titration to trough levels of 5-10 ng/ml
  Interventions: Drug: Everolimus
- Placebo (Placebo Comparator): Placebo treatment for 1 year. Tablets will be identical to everolimus tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Everolimus — Everolimus once daily titrated to trough levels of 5-10 ng/ml.
  Other Names: RAD001; Votubia
  Arms: Everolimus
Drug: Placebo
  Arms: Placebo

SUMMARY:
Tuberous sclerosis complex (TSC) is a genetic disease that leads to mental retardation in over 50% of patients, and to learning problems, behavioral problems, autism and epilepsy in up to 90% of patients. The underlying deficit of TSC, loss of inhibition of the mammalian target of rapamycin (mTOR) protein due to dysfunction of the tuberin/hamartin protein complex, can be rescued by everolimus. Everolimus has been registered as treatment for renal cell carcinoma and giant cell astrocytoma (SEGA). Evidence in human and animal studies suggests that mTOR inhibitors improve learning and development in patients with TSC.

DETAILED DESCRIPTION:
Randomized double-blind placebo controlled intervention study in children with TSC between age 4 and 15 years with an intelligence quotient (IQ) estimated <80 and/or special schooling and/or autism spectrum disorder and/or learning disability requiring remedial teaching.

Patients are randomised to receive everolimus or placebo during a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Children with a definite diagnosis of TSC between 4 and 15 years.
* With an IQ estimated <80 and/or special schooling and/or autism spectrum disorder and/or learning disability requiring remedial teaching.
* Written informed consent by parents/care-takers, and the patient if he or she is 12 years or older and cognitively able to consent.
* In girls after menarche, appropriate contraception must be used or abstinence practiced.

Exclusion Criteria:

* Hepatic dysfunction
* Surgery <6wk
* Current infection at time of inclusion
* Developmental age estimated below 3.5 years
* Intractable epilepsy with more than 1 seizure/week
* Inability to comply with the treatment protocol
* Additional diseases or disorders that may influence the endpoints, including:

  * SEGA requiring treatment
  * Uncontrolled diabetes mellitus
  * Known impaired lung function
* Allergy for any of the components of the study medication
* Prior treatment with mTOR inhibitors
* HIV seropositivity
* Bleeding diathesis or oral anti-vitamin K medication
* Serum creatinine > 1.5 x ULN
* Uncontrolled hyperlipidemia (fasting serum cholesterol > 7.75 mmol/L, fasting serum triglycerides > 2.5 x ULN)
* Use of investigational drug within 30 days prior to inclusion
* History of myocardial infarction, angina or stroke related to atherosclerosis, organ transplantation, malignancy in the past 2 years
* Pregnancy or breastfeeding
* Children at risk for Hepatitis B (HB), unless hepatitis B serology is normal. Risk groups are children who have lived in Asia, Africa, Central and South America, Eastern Europe, Spain, Portugal, and Greece, children with known or suspected past or current hepatitis B infection, current or prior IV illicit drug use, current or prior dialysis, household contact with hepatitis B infected patient(s), current or prior high-risk sexual activity, body piercing or tattoos, mother known to have hepatitis B history. If vaccinated, presence of HBs Ab is normal.
* Known or suspected hepatitis C infection, unless hepatitis C serology is normal.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Cognitive ability measured by IQ | 12 months
  Assessed by Wechsler scales: Wechsler Preschool and Primary Scale of Intelligence (WPPSI-III NL) and Wechsler Intelligence Scale for Children (WISC-III-NL)

SECONDARY OUTCOMES:
Autistic features | 12 Months
  Assessed by Autism Diagnostic Observation Schedule (ADOS)
Social and communicational skills | 12 Months
  Assessed by social responsiveness scale (SRS) and Dutch Children's Communication Checklist (CCC-2-NL) questionnaires
Working memory and attention, information processing | 6 and 12 Months
  Assessed by Cambridge Neuropsychological Test Automated Battery (CANTAB)
Visual-motor integration | 12 Months
  Assessed by BEERY Visual-Motor Integration (BEERY VMI), grooved pegboard
Child behavior | 12 Months
  Assessed by Child Behavior Checklist (CBCL) and Teacher's Report Form (TRF) questionnaires
Executive functioning | 12 Months
  Assessed by Behavior Rating Inventory of Executive Functioning (BRIEF) questionnaire Dutch version
Sleeping problems | 12 Months
  Assessed by Sleep Disturbance Scale for Children (SDSC) questionnaire
Child health | 12 Months
  Assessed by Child Health Questionnaire Parent Form (CHQ-PF50) questionnaire
Sensory related difficulties | 12 Months
  Assessed by Short Sensory Profile (SSP) questionnaire
Epilepsy | 12 Months
  Comparison of epilepsy frequency during month previous to study start and last month of trial participation.
  EEG abnormalities

OTHER OUTCOMES:
School level | 12 Months
  Assessed by the school CITO (centraal instituut voor toetsontwikkeling) scores or reading and arithmetic scores
Pharmacokinetics | 12 Months
  Assessed by measuring trough levels of everolimus
Safety | 12 Months
  Levels of and abnormalities in blood control values

CONTACTS AND LOCATIONS:
Overall Officials: M.C.Y. de Wit, MD. PhD., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

REFERENCES:
- [Derived] Overwater IE, Rietman AB, Mous SE, Bindels-de Heus K, Rizopoulos D, Ten Hoopen LW, van der Vaart T, Jansen FE, Elgersma Y, Moll HA, de Wit MY; ENCORE Expertise Centre for Neurodevelopmental Disorders. A randomized controlled trial with everolimus for IQ and autism in tuberous sclerosis complex. Neurology. 2019 Jul 9;93(2):e200-e209. doi: 10.1212/WNL.0000000000007749. Epub 2019 Jun 19. PMID 31217257